CLINICAL TRIAL: NCT03566810
Title: A Randomized, Open-label, 2-Way-Crossover Study Assessing the Bioequivalence Between Single Doses of 500 mg Glucophage Extended Release (GXR) Tablets (Merck/China Nantong-Manufactured) and 500 mg GXR Tablets (Merck/Germany Darmstadt-Manufactured) Under Fed and Fasted State in Two Groups of Healthy Volunteers
Brief Title: Glucophage Extended Release (GXR) China Bioequivalence Study (Nantong - Darmstadt)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: MS200084_0013
Record Dates: First submitted 2018-06-11; First posted 2018-06-25 (Actual); Results first posted 2020-01-09 (Actual); Last update posted 2020-01-09 (Actual); Status verified 2019-12

CONDITIONS: Healthy
Keywords: Diabetes Mellitus; Glucophage Extended Release (GXR); Bioequivalence Study
MeSH Terms: conditions — Diabetes Mellitus | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- First Test GXR (Fasting), Then Reference GXR (Fasting) (Experimental): Participants received a single oral dose of 500 milligrams (mg) of test GXR tablet (Merck Nantong/China) on Day 1 in treatment period 1 followed by a single oral dose of 500 mg reference GXR (Merck Darmstadt/Germany) on Day 8 in treatment period 2 under fasting conditions. There was a wash-out period of 7 days between each treatment period.
  Interventions: Drug: Test GXR; Drug: Reference GXR
- First Reference GXR (Fasting), Then Test GXR (Fasting) (Experimental): Participants received a single oral dose of 500 mg of reference GXR tablet (Merck Darmstadt/Germany) on Day 1 in treatment period 1 followed by a single oral dose of 500 mg test GXR (Merck Nantong/China) on Day 8 in treatment period 2 under fasting conditions. There was a wash-out period of 7 days between each treatment period.
  Interventions: Drug: Test GXR; Drug: Reference GXR
- First Test GXR (Fed), Then Reference GXR (Fed) (Experimental): Participants received a single oral dose of 500 mg of test GXR tablet (Merck Nantong/China) on Day 1 in treatment period 1 followed by a single oral dose of 500 mg reference GXR (Merck Darmstadt/Germany) on Day 8 in treatment period 2 under fed conditions. There was a wash-out period of 7 days between each treatment period.
  Interventions: Drug: Test GXR; Drug: Reference GXR
- First Reference GXR (Fed), Then Test GXR (Fed) (Experimental): Participants received a single oral dose of 500 mg of reference GXR tablet (Merck Darmstadt/Germany) on Day 1 in treatment period 1 followed by a single oral dose of 500 mg test GXR (Merck Nantong/China) on Day 8 in treatment period 2 under fed conditions. There was a wash-out period of 7 days between each treatment period.
  Interventions: Drug: Test GXR; Drug: Reference GXR

INTERVENTIONS:
Drug: Test GXR — Participants received a single oral dose of 500 mg of test GXR tablet (Merck Nantong/China) under fasting or fed conditions on either Day 1 (Treatment Period 1) or Day 8 (Treatment Period 2).
  Other Names: Metformin hydrochloride
Drug: Reference GXR — Participants received a single oral dose of 500 mg of reference GXR tablet (Merck Darmstadt/France) under fasting or fed conditions on either Day 1 (Treatment Period 1) or Day 8 (Treatment Period 2).
  Other Names: Metformin hydrochloride

SUMMARY:
The study will assess the bioequivalence between single doses of GXR manufactured in Merck Nantong China (test drug) and GXR manufactured in Merck Darmstadt Germany (reference drug) under fed and fasted state in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Overtly healthy as determined by medical evaluation, including medical history and a physical examination
* Have a body weight within 50 to 90 kilogram (kg) and Body mass index (BMI) within the range 18 to 30 kg per meter square (kg/m^2) (inclusive)
* Chinese male and female (at least 1/4 of each gender per study group)
* A male participant must agree to use and to have their female partners use a highly effective contraception (that is, methods with a failure rate of less than 1 percent per year) for a period of at least 1 month before and after dosing
* A female is eligible if she is not pregnant (that is, after a confirmed menstrual period and a negative serum pregnancy test), not breastfeeding, and at least one of the following conditions applies
* Is not a woman of childbearing potential (WOCBP) OR
* Is a WOCBP who agrees to use a highly effective contraceptive method (that is, has a failure rate of less than 1 percent per year) for a period of at least 1 month before and after dosing
* Can give signed informed consent, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and this protocol
* Non-smoker (0 cigarettes, pipes, cigars, or others) since at least 3 months
* All values for biochemistry and hematology tests of blood and urine within the normal range or showing no clinically relevant deviation as judged by the Investigator
* Electrocardiogram recording (12 lead ECG) without signs of clinically relevant pathology as judged by the Investigator.
* Pulse, body temperature, and respiration in sitting position within the normal range or showing no clinically relevant deviation as judged by the Investigator. Blood pressure in sitting position within normal range: greater than or equals to (>=) 90 millimeter of mercury (mmHg) and less than or equal to (=<) 139 mmHg for systolic blood pressure; >= 60 mmHg and =< 90 mmHg for diastolic blood pressure
* Negative screen for alcohol and drugs of abuse (cannabis, benzodiazepines, barbiturates, opiates, cocaine, and methyl amphetamine) at screening and on admission
* Negative screen for hepatitis A virus (HAV) antibodies, hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibodies, human immunodeficiency virus (HIV) antibodies, and Treponema pallidum (TP) antibodies

Exclusion Criteria:

* Participation in a clinical trial within 90 days prior to first drug administration
* Blood donation (equal or more than 500 milliliter [mL]) or significant blood loss within 90 days prior to first drug administration
* Any surgical or medical condition, including findings in the medical history or in the pre-study assessments, or any other significant disease, that in the opinion of the Investigator, constitutes a risk or a contraindication for the participation of the participant in the study or that could interfere with the study objectives, conduct or evaluation
* History of surgery of the gastrointestinal tract which could influence the gastrointestinal absorption and/or motility according to the Investigator's opinion
* History or presence of relevant liver diseases or hepatic dysfunction.
* Allergy: ascertained or presumptive hypersensitivity to the active drug substance and/or formulations' ingredients; history of anaphylaxis to drugs or allergic reactions in general, which the Investigator considers may affect the outcome of the study
* Receipt of any prescription or non-prescription medication within 2 weeks before the first Investigational medicinal product (IMP) administration, including multivitamins and herbal products (that is St John's Wort, or traditional Chinese medicines), except for the permitted medications
* Renal failure or renal dysfunction (creatinine clearance [Ccr] < 80 mL/minute) as assessed by using the estimated measure with the Cockcroft-Gault equation.
* Known lack of participant compliance or inability to communicate or cooperate with the Investigator (example, language problem, poor mental status)
* Non-acceptance of study high-fat breakfast (example, vegetarians, vegans and participants who follow special diets)
* Consumption of large quantities of methylxanthine-containing beverages (>5 cups of coffee/day or equivalent)
* Consumption of grapefruit, cranberry, or juices of these fruits, from 14 days prior to drug administration until collection of the last Pharmacokinetics sample in Period 2
* Any contraindication to Glucophage
* Abnormal and clinically significant chest X-ray finding at screening

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2018-10-11 (Actual); Primary Completion 2018-11-28 (Actual); Study Completion 2018-11-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Pharmaceutical Manufacturing (Jiangsu) Co., Ltd., an affiliate of Merck KGaA, Darmstadt, Germany
Locations (1):
- Xuanwu Hospital Capital Medical University, Beijing, China

RESULTS

PARTICIPANT FLOW:
Groups:
- First Test GXR (Fasting), Then Reference GXR (Fasting): Participants received a single oral dose of 500 milligrams (mg) of test GXR tablet (Merck Nantong, China) on Day 1 in treatment period 1 followed by a single oral dose of 500 mg reference GXR (Merck Darmstadt, Germany) on Day 8 in treatment period 2 under fasting conditions. There was a wash-out period of 7 days between each treatment period.
- First Reference GXR (Fasting), Then Test GXR (Fasting): Participants received a single oral dose of 500 mg of reference GXR tablet (Merck Darmstadt, Germany) on Day 1 in treatment period 1 followed by a single oral dose of 500 mg test GXR (Merck Nantong, China) on Day 8 in treatment period 2 under fasting conditions. There was a wash-out period of 7 days between each treatment period.
- First Test GXR (Fed), Then Reference GXR (Fed): Participants received a single oral dose of 500 mg of test GXR tablet (Merck Nantong, China) on Day 1 in treatment period 1 followed by a single oral dose of 500 mg reference GXR (Merck Darmstadt, Germany) on Day 8 in treatment period 2 under fed conditions. There was a wash-out period of 7 days between each treatment period.
- First Reference GXR (Fed), Then Test GXR (Fed): Participants received a single oral dose of 500 mg of reference GXR tablet (Merck Darmstadt, Germany) on Day 1 in treatment period 1 followed by a single oral dose of 500 mg test GXR (Merck Nantong, China) on Day 8 in treatment period 2 under fed conditions. There was a wash-out period of 7 days between each treatment period.
Period: Treatment Period 1 (Day 1-Day 3)
Arm/Group | First Test GXR (Fasting), Then Reference GXR (Fasting) | First Reference GXR (Fasting), Then Test GXR (Fasting) | First Test GXR (Fed), Then Reference GXR (Fed) | First Reference GXR (Fed), Then Test GXR (Fed)
Started | 19 | 19 | 8 | 8
Treated | 19 | 18 | 8 | 8
Completed | 19 | 18 | 8 | 8
Not Completed | 0 | 1 | 0 | 0
Not completed — Enrolled, but never treated | 0 | 1 | 0 | 0
Period: Treatment Period 2 (Day 8- Day 10)
Arm/Group | First Test GXR (Fasting), Then Reference GXR (Fasting) | First Reference GXR (Fasting), Then Test GXR (Fasting) | First Test GXR (Fed), Then Reference GXR (Fed) | First Reference GXR (Fed), Then Test GXR (Fed)
Started | 19 | 18 | 8 | 8
Completed | 19 | 18 | 8 | 8
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received at least 1 dose of investigational medicinal product (IMP).
Groups:
- Total: Total of all reporting groups
Arm/Group | First Test GXR (Fasting), Then Reference GXR (Fasting) | First Reference GXR (Fasting), Then Test GXR (Fasting) | First Test GXR (Fed), Then Reference GXR (Fed) | First Reference GXR (Fed), Then Test GXR (Fed) | Total
Number analyzed (Participants) | 19 | 18 | 8 | 8 | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.5 (8.00) | 33.5 (8.79) | 32.6 (7.13) | 35.8 (11.15) | 33.0 (8.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 3 | 3 | 19
  Male | 13 | 11 | 5 | 5 | 34
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 19 | 18 | 8 | 8 | 53
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to the Last Sampling Time (AUC 0-t) of Metformin
Description: Area under the plasma concentration versus time curve from time zero to the last sampling time t at which the concentration was at or above the lower limit of quantification (LLQ). AUC0-t was to be calculated according to the mixed log-linear trapezoidal rule.
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 14 post-dose on Day 1 and Day 8; 24, 30, 36 hours post-dose on Day 2 and 9; 48 hours post-dose on Day 3 and 10
Population: The Pharmacokinetic (PK) Analysis Set included all participants who completed the study with adequate study drug compliance, without any relevant protocol violations or events with respect to factors likely to affect comparability of PK results, and with sufficient evaluable data to determine primary outcome measures for both treatments.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*h/mL)
Groups:
- Test GXR (Fasting): Participants received a single oral dose of 500 mg of test GXR tablet (Merck Nantong/China) either on Day 1 in treatment period 1 or on Day 8 in treatment period 2 under fasting conditions.
- Reference GXR (Fasting): Participants received a single oral dose of 500 mg of reference GXR tablet (Merck Darmstadt/France) either on Day 1 in treatment period 1 or on Day 8 in treatment period 2 under fasting conditions.
- Test GXR (Fed): Participants received a single oral dose of 500 mg of test GXR tablet (Merck Nantong/China) either on Day 1 in treatment period 1 or on Day 8 in treatment period 2 under fed conditions.
- Reference GXR (Fed): Participants received a single oral dose of 500 mg of reference GXR tablet (Merck Darmstadt/France) either on Day 1 in treatment period 1 or on Day 8 in treatment period 2 under fed conditions.
Arm/Group | Test GXR (Fasting) | Reference GXR (Fasting) | Test GXR (Fed) | Reference GXR (Fed)
Number analyzed (Participants) | 37 | 37 | 16 | 16
nanogram*hour per milliliter (ng*h/mL) | 3740 (31.5) | 3780 (26.2) | 5500 (17.1) | 5540 (18.7)
Statistical Analysis 1: Comparison: Test GXR (Fasting) vs Reference GXR (Fasting); Statistical Comparison of Test GXR Versus Reference GXR under Fasting conditions; Test type: Equivalence — Analysis was performed with Equivalence Acceptance Range for 90% Confidence Interval (CI) as 80.00% - 125.00%; Ratio of Geometric Least Square(LS)Mean% = 98.69, 90% CI 2-sided [92.20 to 105.64]
Statistical Analysis 2: Comparison: Test GXR (Fed) vs Reference GXR (Fed); Statistical Comparison of Test GXR Versus Reference GXR under Fed conditions; Test type: Equivalence — Analysis was performed with Equivalence Acceptance Range for 90% Confidence Interval (CI) as 80.00% - 125.00%; Ratio of Geometric LS Mean Percentage = 99.39, 90% CI 2-sided [93.15 to 106.05]

2. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Metformin
Description: Pharmacokinetic (PK) parameter Cmax was obtained directly from the concentration versus time curve.
Time Frame: as for outcome 1
Population: The PK Analysis Set included all participants who completed the study with adequate study drug compliance, without any relevant protocol violations or events with respect to factors likely to affect comparability of PK results, and with sufficient evaluable data to determine primary outcome measures for both treatments.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Test GXR (Fasting) | Reference GXR (Fasting) | Test GXR (Fed) | Reference GXR (Fed)
Number analyzed (Participants) | 37 | 37 | 16 | 16
ng/mL | 572 (32.7) | 578 (34.2) | 519 (17.1) | 536 (16.4)
Statistical Analysis 1: Comparison: Test GXR (Fasting) vs Reference GXR (Fasting); Statistical Comparison of Test GXR Versus Reference GXR under Fasting conditions; Test type: Equivalence — Analysis was performed with Equivalence Acceptance Range for 90% Confidence Interval (CI) as 80.00% - 125.00%; Ratio of Geometric LS Mean Percentage = 98.92, 90% CI 2-sided [91.08 to 107.44]
Statistical Analysis 2: Comparison: Test GXR (Fed) vs Reference GXR (Fed); Statistical Comparison of Test GXR Versus Reference GXR under Fed conditions; Test type: Equivalence — Analysis was performed with Equivalence Acceptance Range for 90% Confidence Interval (CI) as 80.00% - 125.00%; Ratio of Geometric LS Mean Percentage = 96.89, 90% CI 2-sided [89.87 to 104.46]

3. Secondary Outcome: Time to Reach Maximum Plasma Concentration of Metformin
Description: Time to reach the maximum plasma concentration (Tmax) was obtained directly from the concentration versus time curve.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Arm/Group | Test GXR (Fasting) | Reference GXR (Fasting) | Test GXR (Fed) | Reference GXR (Fed)
Number analyzed (Participants) | 37 | 37 | 16 | 16
hours | 3.00 [1.00 to 5.00] | 4.00 [1.00 to 5.00] | 6.00 [3.00 to 10.00] | 6.00 [5.00 to 8.00]
Statistical Analysis 1: Comparison: Test GXR (Fasting) vs Reference GXR (Fasting); Statistical Comparison of Test GXR Versus Reference GXR under Fasting conditions; Test type: Equivalence — Analysis was performed with Equivalence Acceptance Range for 90% Confidence Interval (CI) as 80.00% - 125.00%; Median point estimate difference = 0.00, 90% CI 2-sided [-0.50 to 0.00]
Statistical Analysis 2: Comparison: Test GXR (Fed) vs Reference GXR (Fed); Statistical Comparison of Test GXR Versus Reference GXR under Fed conditions; Test type: Equivalence — Analysis was performed with Equivalence Acceptance Range for 90% Confidence Interval (CI) as 80.00% - 125.00%; Median point estimate difference = 0.00, 90% CI 2-sided [-0.50 to 0.50]

4. Secondary Outcome: Apparent Terminal Half-Life (t1/2) of Metformin
Description: Terminal half-life is the time measured for the concentration to decrease by one half. Terminal half-life calculated by natural log 2 divided by lambda z.
Time Frame: as for outcome 1
Population: The Pharmacokinetic analysis set. Here "Number of participants analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Test GXR (Fasting) | Reference GXR (Fasting) | Test GXR (Fed) | Reference GXR (Fed)
Number analyzed (Participants) | 37 | 35 | 16 | 15
hours | 5.80 (63.7) | 5.56 (58.4) | 5.34 (65.1) | 5.37 (99.8)

5. Secondary Outcome: Area Under the Plasma Concentration-Time Curve From Time 0 to Infinity (AUC0-inf) of Metformin
Description: AUC0-inf was calculated by combining AUC0-t and AUCextra. AUC extra represents an extrapolated value obtained by Clast/ lambda z, where Clast is the calculated plasma concentration at the last sampling time point at which the measured plasma concentration is at or above the Lower Limit of quantification (LLQ) and lambda z is the apparent terminal rate constant determined by log-linear regression analysis of the measured plasma concentrations of the terminal log-linear phase.
Time Frame: as for outcome 1
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Test GXR (Fasting) | Reference GXR (Fasting) | Test GXR (Fed) | Reference GXR (Fed)
Number analyzed (Participants) | 37 | 35 | 16 | 15
ng*h/mL | 3890 (29.4) | 3980 (25.0) | 5630 (17.2) | 5750 (19.2)
Statistical Analysis 1: Comparison: Test GXR (Fasting) vs Reference GXR (Fasting); Statistical Comparison of Test GXR Versus Reference GXR under Fasting conditions; Test type: Equivalence — Analysis was performed with Equivalence Acceptance Range for 90% Confidence Interval (CI) as 80.00% - 125.00%; Ratio of Geometric LS Mean Percentage = 97.89, 90% CI 2-sided [91.38 to 104.86]
Statistical Analysis 2: Comparison: Test GXR (Fed) vs Reference GXR (Fed); Statistical Comparison of Test GXR Versus Reference GXR under Fed conditions; Test type: Equivalence — Analysis was performed with Equivalence Acceptance Range for 90% Confidence Interval (CI) as 80.00% - 125.00%; Ratio of Geometric LS Mean Percentage = 98.08, 90% CI 2-sided [92.37 to 104.14]

6. Secondary Outcome: Area Under the Plasma Concentration-Time Curve From Time Tlast Extrapolated to Infinity (AUCextra) of Metformin
Description: AUCextra% was defined as area under the curve from time tlast extrapolated to infinity as percentage of AUC 0-infinity. Here, tlast is the last sampling time at which the concentration is at or above the lower limit of quantification.
Time Frame: as for outcome 1
Population: As AUCextra was >20% of AUC0-inf, parameters derived from lambda z including AUCextra% were regarded as unreliable estimate of the extent of exposure and not calculated as it was pre-specified to not report these data in this condition.
Arm/Group | Test GXR (Fasting) | Reference GXR (Fasting) | Test GXR (Fed) | Reference GXR (Fed)
Number analyzed (Participants) | 0 | 0 | 0 | 0

7. Secondary Outcome: Elimination Rate Constant (Lambda z) of Metformin
Description: Lambda z was determined from the terminal slope of the log-transformed plasma concentration curve using linear regression method.
Time Frame: as for outcome 1
Population: As AUCextra was >20% of AUC0-inf, parameters derived from lambda z were regarded as unreliable estimate of the extent of exposure and not calculated as it was pre-specified to not report these data in this condition.
Arm/Group | Test GXR (Fasting) | Reference GXR (Fasting) | Test GXR (Fed) | Reference GXR (Fed)
Number analyzed (Participants) | 0 | 0 | 0 | 0

8. Secondary Outcome: Total Body Clearance (CL/f) of Metformin
Description: Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes.
Time Frame: as for outcome 1
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter per hour
Arm/Group | Test GXR (Fasting) | Reference GXR (Fasting) | Test GXR (Fed) | Reference GXR (Fed)
Number analyzed (Participants) | 37 | 35 | 16 | 15
liter per hour | 128 (29.4) | 126 (25.0) | 88.9 (17.2) | 87.0 (19.2)

9. Secondary Outcome: Apparent Volume of Distribution at After Extravascular Administration (Vz/f) of Metformin
Description: Vz/f is defined as the distribution of a study drug between plasma and the rest of the body after oral dosing.
Time Frame: as for outcome 1
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter
Arm/Group | Test GXR (Fasting) | Reference GXR (Fasting) | Test GXR (Fed) | Reference GXR (Fed)
Number analyzed (Participants) | 37 | 35 | 16 | 15
liter | 1070 (75.6) | 1010 (61.1) | 684 (65.8) | 674 (93.7)

10. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious TEAEs
Description: An Adverse event (AE) was defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease associated with the use of study drug, whether or not considered related to the study drug or worsening of pre-existing medical condition, whether or not related to study drug. A serious adverse event (SAE) was an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. An AE was considered as 'treatment emergent' if it occurred after the first drug administration of each period or if it was present prior to drug administration but exacerbated after the drug administration. TEAEs included both Serious TEAEs and non-serious TEAEs.
Time Frame: Time from informed consent up to end of study (Day 15)
Population: The Safety Analysis Set included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Test GXR (Fasting) | Reference GXR (Fasting) | Test GXR (Fed) | Reference GXR (Fed)
Number analyzed (Participants) | 37 | 37 | 16 | 16
Participants
  TEAEs | 10 | 11 | 3 | 4
  Serious TEAEs | 0 | 0 | 0 | 0

11. Secondary Outcome: Number of Participants With Clinically Significant Abnormalities in Vital Signs
Description: Vital sign assessment included blood pressure, pulse rate, body temperature and respiration (frequency per minute). Number of participants with clinically significant abnormalities in vital signs were reported. Clinically significance was decided by investigator.
Time Frame: Time from informed consent up to end of study (Day 15)
Population: The Safety Analysis Set included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Test GXR (Fasting) | Reference GXR (Fasting) | Test GXR (Fed) | Reference GXR (Fed)
Number analyzed (Participants) | 37 | 37 | 16 | 16
Participants | 0 | 0 | 0 | 0

12. Secondary Outcome: Number of Participants With Clinically Significant Abnormalities in Laboratory Values
Description: The laboratory measurements included hematology, blood chemistry and urinalysis. Number of participants with clinically significant abnormalities in laboratory values were reported. Clinically Significance was decided by investigator.
Time Frame: Time from informed consent up to end of study (Day 15)
Population: The Safety Analysis Set included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Test GXR (Fasting) | Reference GXR (Fasting) | Test GXR (Fed) | Reference GXR (Fed)
Number analyzed (Participants) | 37 | 37 | 16 | 16
Participants | 0 | 0 | 0 | 0

13. Secondary Outcome: Number of Participants With Clinically Significant Abnormalities in Physical Examination Findings
Description: Physical examination included assessments of the general appearance, skin and mucosa, superficial lymph nodes, head and neck, chest, abdomen, musculoskeletal, and neurological systems. Number of participants with clinically significant abnormalities in physical examination findings were reported. clinically significance was decided by investigator.
Time Frame: Time from informed consent up to end of study (Day 15)
Population: The Safety Analysis Set included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Test GXR (Fasting) | Reference GXR (Fasting) | Test GXR (Fed) | Reference GXR (Fed)
Number analyzed (Participants) | 37 | 37 | 16 | 16
Participants | 0 | 0 | 0 | 0

14. Secondary Outcome: Number of Participants With Clinically Significant Abnormalities in 12-lead Electrocardiogram (ECG) Findings
Description: The 12-lead ECG recordings were obtained after 5 minutes of rest in a semi-supine position. ECG recordings included rhythm, ventricular rate, PR interval, QRS duration, QT and QTc intervals. Number of participants with clinically significant abnormalities in 12-lead ECG findings were reported. Clinically significance was decided by investigator.
Time Frame: Time from informed consent up to end of study (Day 15)
Population: The Safety Analysis Set included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Test GXR (Fasting) | Reference GXR (Fasting) | Test GXR (Fed) | Reference GXR (Fed)
Number analyzed (Participants) | 37 | 37 | 16 | 16
Participants | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Time from informed consent up to end of study (Day 15)
Description: The Safety Analysis Set included all participants who received at least 1 dose of study drug.
Arm/Group | Test GXR (Fasting) | Reference GXR (Fasting) | Test GXR (Fed) | Reference GXR (Fed)
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/37 | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/37 | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 10/37 | 11/37 | 3/16 | 4/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Test GXR (Fasting) (N=37) | Reference GXR (Fasting) (N=37) | Test GXR (Fed) (N=16) | Reference GXR (Fed) (N=16)
Diarrhoea (Gastrointestinal disorders) | 8 | 6 | 1 | 3
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 3 | 0 | 0
Furuncle (Infections and infestations) | 1 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 1
White blood cell count decreased (Investigations) | 1 | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 0 | 0 | 0
Electrocardiogram ST segment abnormal (Investigations) | 0 | 0 | 1 | 0
Chest pain (General disorders) | 0 | 1 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-04-19): https://cdn.clinicaltrials.gov/large-docs/10/NCT03566810/Prot_000.pdf
  • Statistical Analysis Plan (2018-12-20): https://cdn.clinicaltrials.gov/large-docs/10/NCT03566810/SAP_001.pdf